CLINICAL TRIAL: NCT02204540
Title: Validation of Video Monitoring to Assess Compliance in Clinical Interventions
Brief Title: Feasibility of Using Webcams in Clinical Studies
Acronym: WEBCAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Courtney Peterson, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PBRC 2014-033
Record Dates: First submitted 2014-07-27; First posted 2014-07-30 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Video Monitoring Via Webcams
Keywords: Webcams, video monitoring, compliance, adherence
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitoring by webcam (Experimental): Participants will perform a task for a mock clinical study (e.g., swallowing a pill, consuming food) while being recorded and monitored by webcam.
  Interventions: Behavioral: Mock study intervention
- In-person monitoring (Active Comparator): Participants will perform a task for a mock clinical study (e.g., swallowing a pill, consuming good) while being monitored in-person.
  Interventions: Behavioral: Mock study intervention

INTERVENTIONS:
Behavioral: Mock study intervention — Participants will swallow a pill and consume food in a mock research study, while their performance of the task is being monitored.

SUMMARY:
This study tests the feasibility of having study participants use webcams to participate in research studies. The study scientists hypothesize (1) that webcams will be an adequate method of detecting a participant's ability to perform a tasks for a clinical trial (e.g., swallowing a pill, eating food) and (2) that a majority of study participants would be willing to use a webcam to participate in a research study.

DETAILED DESCRIPTION:
In the first phase of this study, the study scientists will research and compare technologies that will be used in video monitoring via webcam. The study team will also develop a standardized protocol for using the webcam technology through hands-on testing (without the use of study participants).

In the second phase of this study, video monitoring via webcam will be tested. Specifically, the study scientists will see whether the video recordings can be used to assess compliance to clinical interventions. Study participants will be recruited from among Pennington Biomedical Research Center employees and assigned to be either evaluators or testers. Testers will act as if they were study participants in a clinical study who are supposed to adhere to an intervention such as swallowing a pill or consuming food. They will be video-recorded by webcam while performing these tasks. Evaluators will then try to detect how well the testers followed the instructions for the task through in-person observation and by watching video recordings. Data from these tests will then be used to see whether watching the video recordings is as effective as watching in-person.

In the third phase of this study, past, current, and potential study participants at Pennington Biomedical Research Center will be surveyed to determine their comfort with using webcams and their likeliness to opt to use webcams to participate in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Pennington Biomedical Research Center employees and trainees
* Age 18 years and older

Exclusion Criteria:

* Any employees who directly report to and are directly employed by the study's principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity of Detecting Non-Compliance | 1 Month
  The sensitivity (true positive rate, as a percentage of total non-compliant events) of observers charged with detecting non-compliance to a mock study intervention will be tested both via in-person monitoring and monitoring by webcam. The mock study interventions that will be monitored will include pill swallowing and eating. Non-compliance events will be chosen from a defined list of non-compliant behaviors (e.g., tampering with the pill, spitting food into a napkin and not eating it), and will be performed by mock study participants. The observers will record the number of non-compliant events they actually observe the mock study participants performing. This data will be analyzed as described here in order to determine the validity of monitoring non-compliance by webcam, in comparison to in-person monitoring.

SECONDARY OUTCOMES:
Specificity and Inter-Rater Agreement of Detecting Non-Compliance | 1 Month
  The specificity (false positive rate, as a percentage of distinct events) and inter-rater agreement (as a percentage of total events and as calculated via Cohen's kappa) of observers who are charged with monitoring and recording non-compliance events in-person versus by webcam will also be assessed, similarly as described above.
Attitudes Towards Using Webcams To Participate in Clinical Interventions | 1 year
  A survey will be given to determine potential and current study participants' comfort with video recording technologies and assess their likeliness to opt to use webcams to participate in a clinical study.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney M Peterson, PhD, MSc, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States